CLINICAL TRIAL: NCT01560039
Title: Voluntary Modulation of M1 Motor Cortex Activity Using EEG Neurofeedback for the Treatment of Resistant Chronic Neuropathic Pain - a Clinical and fMRI Study
Brief Title: Electroencephalography Based Neurofeedback in Chronic Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMS-12-HS-0577-11-TLV-CTIL
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; neurostimulation
MeSH Terms: conditions — Neuralgia | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Real EEG-NF (Active Comparator): 10 EEG based neurofeedback sessions modulating the activity of the primary motor cortex
  Interventions: Other: Neurofeedback
- Sham EEG-NF (Sham Comparator): 10 sessions of Sham EEG_NF of the motor cortex area
  Interventions: Other: Sham neurofeedback
- Transcrainal Magnetic Stimulation (Active Comparator): 10 dailt TMS stimulation sessions of M1
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial magentic stimulation of the motor cortex. Device Details : Model is Magstim TMS Rapid. Manufacturer : MAGSTIM CO LTD. Spring Gardens, Whitland, Carmarthenshire, Wales, U.K., SA34 0HR
  Arms: Transcrainal Magnetic Stimulation
Other: Neurofeedback — EEG neurofeedback based on the primary motor cortex
  Arms: Real EEG-NF
Other: Sham neurofeedback — Sham EEG neurofeedback
  Arms: Sham EEG-NF

SUMMARY:
Chronic neuropathic pain is a global health concern, affecting millions of patients worldwide. It is often extremely debilitating and poses a diagnostic and therapeutic challenge. The current mainstay of treatment is pharmacotherapy consisting of powerful analgesics combined with different classes of drugs that change nerve cell membrane properties. However, response to pharmacotherapy is often poor and mandates interventional strategies. Among the latest and most promising interventional strategies is the use of neurostimulation to targeted brain areas, specifically the primary motor cortex . Motor cortex stimulation , both invasive and noninvasive (using megnetic or electical stimulation), has emerged as a highly beneficial treatment, and is currently included in different professional guidelines for the treatment of medically refractory neuropathic pain.

A possible alternative way to achieve stimulation of the motor cortex is by using EEG based neurofeedback. This design, which is actually a Brain Computer Interface (BCI) enables the patient to voluntarily modulate the activity of a circumscribed brain area after a few training sessions. While EEG based neurofeedfback is decades old, it has never been tested in neuropathic pain patients.

This experiment is intended to compare both the clinical effects and the brain correlates of a BCI based self modulation of M1 activity and of exogenous magnetic brain stimulation in a population of patients suffering from chronic neuropathic pain of an upper limb. 15 such patients will receive a course of 10 daily magnetic stimulation sessions with stimulation of M1 as described in the literature. A further 30 patients will be divided into two groups: 15 will perform a course of 10 real BCI neurofeedback sessions modulating motor cortex activity and 15 will perform a course of 10 sham neurofeedback sessions. The participants' baseline chronic pain levels and their response to acute painful stimuli will be clinically evaluated before and after the course, and for an additional 1 month. Furthermore, before and after the course patients will be scanned using functional MRI during rest (baseline pain levels) and during acute pain. These scans are performed both to describe the neural correlates of the analgesia induced by motor cortex magnetic stimulation , and to compare the observed networks to the network effect of a BCI neurofeedback modulation of motor cortex activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, treated medically for neuropathic pain of an upper arm with unsatisfactory results (average daily VAS score over 4)

Exclusion Criteria:

* Cognitive decline,
* malignant disease,
* focal neurological deficit,
* illegal substance abuse
* noncompliance with medical therapy or follow up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
daily pain levels | during three weeks of treatments
  daily pain levels will be assessed using a visual assessment score (VAS) during the treament phase (lasting aproximately 3 weeks)

SECONDARY OUTCOMES:
Daily pain measures for one month following the last session | one month following the last treatment session
  Daily pain scores based on the VAS (visual-analogue scale) system will be assessed for a further one month following the last treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, MD, PhD, Study Director — Sourasky Medical Center
Locations (1):
- Functional Brain Center, Sourasky Medical Center, Tel Aviv, Israel